CLINICAL TRIAL: NCT05002478
Title: Short-Term Effect of Prone Positioning in Infants with Severe Acute Respiratory Distress Syndrome
Brief Title: Infants with Severe Acute Respiratory Distress Syndrome: the Prone Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Tobias Werther, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1426/2021
Record Dates: First submitted 2021-07-29; First posted 2021-08-12 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS); Surfactant Dysfunction; Infant
Keywords: Acute Respiratory Distress Syndrome; Electrical Impedance Tomography; Lung Ultrasonography; Prone Position; Infants
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Surfactant Dysfunction | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: Single center randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prone Group (Experimental): Turn patient in prone position after surfactant administration. After 6 hours turn patient in supine position and perform EIT and LUS.
  Interventions: Other: Prone positioning
- Supine Group (No Intervention): Leave patient in supine position after surfactant administration. After 6 hours perform EIT and LUS.

INTERVENTIONS:
Other: Prone positioning — Turn patient in prone position after surfactant administration.
  Arms: Prone Group

SUMMARY:
The main objective is to determine the short-term effect of prone positioning in infants with infection-associated severe acute respiratory distress syndrome. The investigators compare oxygenation parameters and measurements from electrical impedance tomography (EIT) and lung ultrasonography (LUS) in mechanically ventilated infants in prone position versus supine position after surfactant administration.

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) is an acute lung injury that can be triggered by pulmonary (direct lung injury) and extrapulmonary (indirect lung injury) etiologies. Pediatric ARDS (pARDS) occurs in approximately 3% of children admitted to intensive care units (ICUs) and is associated with approximately 17% mortality. The primary etiologies of pARDS have been summarized as pneumonia (35%), aspiration (15%), sepsis (13%), near-drowning (9%), cardiac disease (7%), and other clinical conditions (21%). ARDS manifests as pulmonary inflammation, alveolar edema, and hypoxemic respiratory failure. Mechanical ventilation remains an essential component in the care of patients with ARDS. Many adjunctive treatments rely on pathophysiological considerations. The pathophysiology of ARDS is characterized by inflammatory, proliferative, and fibrotic phases. The different phases induce a ventilation-perfusion mismatch. Inflammation causes surfactant inactivation and depletion. A number of clinical studies have reported clinical benefits following the instillation of exogenous surfactant in pediatric patients with acute respiratory failure. On the other side, prone positioning seem to be a promising intervention in critically ill infants and children with infection-associated acute lung injury. However, data conflict on the use of prone positioning in pediatric patients with acute lung injury.

Turning patients with moderate to severe lung disease into prone position has shown many positive effects. Prolonged intervals of prone positioning have been associated with a decrease in mortality in adult patients with acute respiratory failure. An increase in partial pressure of oxygen (PaO2)/fraction of inspired oxygen (FiO2) has been described after 4 hours in prone position in adult patients with severe acute respiratory failure. Similarly, a decrease of the oxygenation index has been found after 8 hours of prone positioning in adult patients with respiratory failure from coronavirus disease of 2019 (COVID-19) associated acute respiratory distress syndrome. The process of prone positioning appeared safe also in critically ill infants and children. In a randomized control trial, it has been shown that in 90% of prone positioning oxygenation index decreased of more than 10% in children with acute lung injury.

Electrical impedance tomography (EIT) and lung ultrasound (LUS) are two non-invasive methods to monitor aeration and lung function parameters. EIT can quantify regional distribution of ventilation as well as improvement in end-expiratory air content. EIT has been used at bedside in critically ill adult patients to measure effects of prone position and also in infants with respiratory distress syndrome. On the other side, LUS has become an increasingly popular diagnostic bedside tool for lung examination. It is considered reliable and fast to detect various lung-related pathologies, such as pneumonia, atelectasis, pneumothorax, and interstitial syndrome.

The main objective is to determine the short-term effect of prone positioning in infants with infection-associated severe acute respiratory distress syndrome. To accomplish this, oxygenation parameters and measurements from EIT and LUS will be compared in mechanically ventilated infants in prone position versus supine position after surfactant administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized at Pediatric Intensive Care Unit (PICU) or Neonatal Intensive Care Unit (NICU) of the Medical University Vienna.
* Patients aged >36 weeks (corrected gestational age) and <24 months.
* Patient intubated and mechanically ventilated for at least 6 hours, with an expected requirement of invasive ventilatory support for at least 12 hours.
* Clinical picture strongly suggestive for acute bronchiolitis or pneumonia (fever, fine crackles, prolonged expiration, lung hyperinflation and/or findings of new infiltrates consistent with acute pulmonary parenchymal disease on chest X-ray).
* Severe pediatric acute respiratory distress syndrome (ARDS), defined by OSI ≥12.3 (wean FIO2 to maintain SpO2 ≤ 97% to calculate oxygen saturation index).
* Written informed consent obtained from parents.

Exclusion Criteria:

* Clinical context

  * Need for O2 supplementation to maintain SpO2>94% in the 4 weeks preceding hospitalization in the PICU/NICU
  * Cyanotic congenital heart disease Cardiogenic pulmonary edema
  * Severe pulmonary hypertension
  * Untreated pneumothorax
  * Severe neurological abnormalities
  * Other severe congenital anomalies such as congenital diaphragmatic hernia
  * Ongoing cardiopulmonary resuscitation or limitation of life support
* Contradictions for prone positioning (adapted from Guerin, C., et al., Prone positioning in severe acute respiratory distress syndrome. N Engl J Med, 2013. 368(23): p. 2159-68):

  * Intracranial pressure >30 millimeters of mercury (mmHg) in supine position or cerebral perfusion pressure <60 mmHg
  * Massive hemoptysis requiring an immediate surgical or interventional radiology procedure
  * Tracheal surgery or sternotomy during the previous 15 days
  * Serious facial trauma or facial surgery during the previous 15 days
  * Deep venous thrombosis treated for less than 2 days
  * Cardiac pacemaker inserted in the last 2 days
  * Unstable spine, femur, or pelvic fractures
  * Use of extracorporeal membrane oxygenation (ECMO) before inclusion
  * Lung transplantation
  * Burns on more than 20% of the body surface
* Other non-inclusion criteria

  * Indication not to attempt resuscitation
  * Patient already recruited for other clinical studies
  * Patients who already received surfactant in the last 4 weeks
  * Thoracic skin lesions or wounds on the thorax, where the EIT-electrode-belt would be placed

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Oxygenation saturation index | Change from baseline oxygenation saturation index at 6 hours
  Oxygenation saturation index (OSI) defined by [FiO2 x mean airway pressure x 100]/Peripheral oxygen saturation (SpO2) in millibar [mbar] (wean FiO2 to maintain SpO2 ≤ 97% to calculate OSI).
  OSI values will be calculated after a stable value of SpO2 and mean airway pressure (MAP) will be reached (see ventilation management). The OSI gradient will be calculated as follows: 100*((OSI (0) - OSI (6h)) / OSI (0) = change of OSI in %. OSI (0) accounts for the OSI prior to the prone position (intervention) and OSI (6h) accounts for the OSI six hours after the intervention.

SECONDARY OUTCOMES:
Chang in Lung Ultrasound | Change from baseline LUS score at 6 hours
  Each lung (left and right) is divided into 6 areas (upper anterior, lower anterior, upper lateral, lower lateral, upper posterior, lower posterior). The Lung Ultrasound Score is assigned as follows: 0 indicates A-pattern (defined by the presence of the only A-lines); 1, B-pattern (defined as the presence of ≥3 well-spaced B-lines); 2, severe B pattern (defined as the presence of crowded and coalescent B-lines with or without consolidations limited to the subpleural space); and 3, extended consolidations. The total LUS score ranges from 0 (best) to 36.
Change in the Distribution of the End-Expiratory Lung Volume | Change from baseline EELV at 6 hours
  End-expiratory lung impedance (EELV) is the average of the measured impedance at the end of expiration [arbitrary units].
Change in the Distribution of the Tidal Volume | Change from baseline tidal volume at 6 hours
  Tidal volume is the average difference of end-inspiratory and end-expiratory impedance measurements [arbitrary units].

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Werther, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheifetz IM. Pediatric ARDS. Respir Care. 2017 Jun;62(6):718-731. doi: 10.4187/respcare.05591. PMID 28546374
- [Background] Khemani RG, Smith L, Lopez-Fernandez YM, Kwok J, Morzov R, Klein MJ, Yehya N, Willson D, Kneyber MCJ, Lillie J, Fernandez A, Newth CJL, Jouvet P, Thomas NJ; Pediatric Acute Respiratory Distress syndrome Incidence and Epidemiology (PARDIE) Investigators; Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Paediatric acute respiratory distress syndrome incidence and epidemiology (PARDIE): an international, observational study. Lancet Respir Med. 2019 Feb;7(2):115-128. doi: 10.1016/S2213-2600(18)30344-8. Epub 2018 Oct 22. PMID 30361119
- [Background] Santschi M, Randolph AG, Rimensberger PC, Jouvet P; Pediatric Acute Lung Injury Mechanical Ventilation Investigators; Pediatric Acute Lung Injury and Sepsis Investigators Network; European Society of Pediatric and Neonatal Intensive Care. Mechanical ventilation strategies in children with acute lung injury: a survey on stated practice pattern*. Pediatr Crit Care Med. 2013 Sep;14(7):e332-7. doi: 10.1097/PCC.0b013e31828a89a2. PMID 23842587
- [Background] Orloff KE, Turner DA, Rehder KJ. The Current State of Pediatric Acute Respiratory Distress Syndrome. Pediatr Allergy Immunol Pulmonol. 2019 Jun 1;32(2):35-44. doi: 10.1089/ped.2019.0999. Epub 2019 Jun 17. PMID 31236307
- [Background] Mok YH, Lee JH, Rehder KJ, Turner DA. Adjunctive treatments in pediatric acute respiratory distress syndrome. Expert Rev Respir Med. 2014 Dec;8(6):703-16. doi: 10.1586/17476348.2014.948854. Epub 2014 Aug 13. PMID 25119574
- [Background] Gattinoni L, Taccone P, Carlesso E, Marini JJ. Prone position in acute respiratory distress syndrome. Rationale, indications, and limits. Am J Respir Crit Care Med. 2013 Dec 1;188(11):1286-93. doi: 10.1164/rccm.201308-1532CI. PMID 24134414
- [Background] De Luca D, Cogo P, Kneyber MC, Biban P, Semple MG, Perez-Gil J, Conti G, Tissieres P, Rimensberger PC. Surfactant therapies for pediatric and neonatal ARDS: ESPNIC expert consensus opinion for future research steps. Crit Care. 2021 Feb 22;25(1):75. doi: 10.1186/s13054-021-03489-6. PMID 33618742
- [Background] Amigoni A, Pettenazzo A, Stritoni V, Circelli M. Erratum to: Surfactants in Acute Respiratory Distress Syndrome in Infants and Children: Past, Present and Future. Clin Drug Investig. 2017 Jul;37(7):711. doi: 10.1007/s40261-017-0544-x. No abstract available. PMID 28589372
- [Background] Luchetti M, Ferrero F, Gallini C, Natale A, Pigna A, Tortorolo L, Marraro G. Multicenter, randomized, controlled study of porcine surfactant in severe respiratory syncytial virus-induced respiratory failure. Pediatr Crit Care Med. 2002 Jul;3(3):261-268. doi: 10.1097/00130478-200207000-00011. PMID 12780967
- [Background] Jat KR, Chawla D. Surfactant therapy for bronchiolitis in critically ill infants. Cochrane Database Syst Rev. 2015 Aug 24;2015(8):CD009194. doi: 10.1002/14651858.CD009194.pub3. PMID 26299681
- [Background] Willson DF, Thomas NJ, Markovitz BP, Bauman LA, DiCarlo JV, Pon S, Jacobs BR, Jefferson LS, Conaway MR, Egan EA; Pediatric Acute Lung Injury and Sepsis Investigators. Effect of exogenous surfactant (calfactant) in pediatric acute lung injury: a randomized controlled trial. JAMA. 2005 Jan 26;293(4):470-6. doi: 10.1001/jama.293.4.470. PMID 15671432
- [Background] Ward NS. Effects of prone position ventilation in ARDS. An evidence-based review of the literature. Crit Care Clin. 2002 Jan;18(1):35-44. doi: 10.1016/s0749-0704(03)00063-0. PMID 11910731
- [Background] Lupton-Smith A, Argent A, Rimensberger P, Frerichs I, Morrow B. Prone Positioning Improves Ventilation Homogeneity in Children With Acute Respiratory Distress Syndrome. Pediatr Crit Care Med. 2017 May;18(5):e229-e234. doi: 10.1097/PCC.0000000000001145. PMID 28328787
- [Background] Sud S, Friedrich JO, Taccone P, Polli F, Adhikari NK, Latini R, Pesenti A, Guerin C, Mancebo J, Curley MA, Fernandez R, Chan MC, Beuret P, Voggenreiter G, Sud M, Tognoni G, Gattinoni L. Prone ventilation reduces mortality in patients with acute respiratory failure and severe hypoxemia: systematic review and meta-analysis. Intensive Care Med. 2010 Apr;36(4):585-99. doi: 10.1007/s00134-009-1748-1. Epub 2010 Feb 4. PMID 20130832
- [Background] Curley MA, Hibberd PL, Fineman LD, Wypij D, Shih MC, Thompson JE, Grant MJ, Barr FE, Cvijanovich NZ, Sorce L, Luckett PM, Matthay MA, Arnold JH. Effect of prone positioning on clinical outcomes in children with acute lung injury: a randomized controlled trial. JAMA. 2005 Jul 13;294(2):229-37. doi: 10.1001/jama.294.2.229. PMID 16014597
- [Background] Munshi L, Del Sorbo L, Adhikari NKJ, Hodgson CL, Wunsch H, Meade MO, Uleryk E, Mancebo J, Pesenti A, Ranieri VM, Fan E. Prone Position for Acute Respiratory Distress Syndrome. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2017 Oct;14(Supplement_4):S280-S288. doi: 10.1513/AnnalsATS.201704-343OT. PMID 29068269
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Chatte G, Sab JM, Dubois JM, Sirodot M, Gaussorgues P, Robert D. Prone position in mechanically ventilated patients with severe acute respiratory failure. Am J Respir Crit Care Med. 1997 Feb;155(2):473-8. doi: 10.1164/ajrccm.155.2.9032181.
- [Background] Mittermaier M, Pickerodt P, Kurth F, de Jarcy LB, Uhrig A, Garcia C, Machleidt F, Pergantis P, Weber S, Li Y, Breitbart A, Bremer F, Knape P, Dewey M, Doellinger F, Weber-Carstens S, Slutsky AS, Kuebler WM, Suttorp N, Muller-Redetzky H. Evaluation of PEEP and prone positioning in early COVID-19 ARDS. EClinicalMedicine. 2020 Nov;28:100579. doi: 10.1016/j.eclinm.2020.100579. Epub 2020 Oct 11. PMID 33073217
- [Background] Fineman LD, LaBrecque MA, Shih MC, Curley MA. Prone positioning can be safely performed in critically ill infants and children. Pediatr Crit Care Med. 2006 Sep;7(5):413-22. doi: 10.1097/01.PCC.0000235263.86365.B3. PMID 16885792
- [Background] Baudin F, Emeriaud G, Essouri S, Beck J, Portefaix A, Javouhey E, Guerin C. Physiological Effect of Prone Position in Children with Severe Bronchiolitis: A Randomized Cross-Over Study (BRONCHIO-DV). J Pediatr. 2019 Feb;205:112-119.e4. doi: 10.1016/j.jpeds.2018.09.066. Epub 2018 Nov 14. PMID 30448014
- [Background] Becher T, Kott M, Schadler D, Vogt B, Meinel T, Weiler N, Frerichs I. Influence of tidal volume on ventilation inhomogeneity assessed by electrical impedance tomography during controlled mechanical ventilation. Physiol Meas. 2015 Jun;36(6):1137-46. doi: 10.1088/0967-3334/36/6/1137. Epub 2015 May 26. PMID 26007294
- [Background] Dalla Corte F, Mauri T, Spinelli E, Lazzeri M, Turrini C, Albanese M, Abbruzzese C, Lissoni A, Galazzi A, Eronia N, Bronco A, Maffezzini E, Pesenti A, Foti G, Bellani G, Grasselli G. Dynamic bedside assessment of the physiologic effects of prone position in acute respiratory distress syndrome patients by electrical impedance tomography. Minerva Anestesiol. 2020 Oct;86(10):1057-1064. doi: 10.23736/S0375-9393.20.14130-0. Epub 2020 May 22. PMID 32449339
- [Background] Corsini I, Parri N, Ficial B, Dani C. Lung ultrasound in the neonatal intensive care unit: Review of the literature and future perspectives. Pediatr Pulmonol. 2020 Jul;55(7):1550-1562. doi: 10.1002/ppul.24792. Epub 2020 Apr 27. PMID 32339409
- [Background] Khemani RG, Smith LS, Zimmerman JJ, Erickson S; Pediatric Acute Lung Injury Consensus Conference Group. Pediatric acute respiratory distress syndrome: definition, incidence, and epidemiology: proceedings from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med. 2015 Jun;16(5 Suppl 1):S23-40. doi: 10.1097/PCC.0000000000000432. PMID 26035358
- [Background] Curley MA, Arnold JH, Thompson JE, Fackler JC, Grant MJ, Fineman LD, Cvijanovich N, Barr FE, Molitor-Kirsch S, Steinhorn DM, Matthay MA, Hibberd PL; Pediatric Prone Positioning Study Group. Clinical trial design--effect of prone positioning on clinical outcomes in infants and children with acute respiratory distress syndrome. J Crit Care. 2006 Mar;21(1):23-32; discussion 32-7. doi: 10.1016/j.jcrc.2005.12.004. PMID 16616620
- [Background] Rey-Santano C, Mielgo VE, Andres L, Ruiz-del-Yerro E, Valls-i-Soler A, Murgia X. Acute and sustained effects of aerosolized vs. bolus surfactant therapy in premature lambs with respiratory distress syndrome. Pediatr Res. 2013 May;73(5):639-46. doi: 10.1038/pr.2013.24. Epub 2013 Feb 12. PMID 23403804
- [Background] Bianco F, Ricci F, Catozzi C, Murgia X, Schlun M, Bucholski A, Hetzer U, Bonelli S, Lombardini M, Pasini E, Nutini M, Pertile M, Minocchieri S, Simonato M, Rosa B, Pieraccini G, Moneti G, Lorenzini L, Catinella S, Villetti G, Civelli M, Pioselli B, Cogo P, Carnielli V, Dani C, Salomone F. From bench to bedside: in vitro and in vivo evaluation of a neonate-focused nebulized surfactant delivery strategy. Respir Res. 2019 Jul 2;20(1):134. doi: 10.1186/s12931-019-1096-9. PMID 31266508